CLINICAL TRIAL: NCT03729752
Title: PET Imaging of Radiolabeled Anti-HIV-1 Envelope Monoclonal Antibody (VRC01)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Principal Investigator, Timothy Henrich, Associate Professor of Medicine, University of California, San Francisco
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-23507
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: HIV-1-infection
Keywords: HIV-1-infection; PET scan; MRI; Viremia; Antiretroviral therapy
MeSH Terms: conditions — Viremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteer (Active Comparator): Four serial PET-MR scans over 120 hours following a single, bolus injection of [89]Zr-DFO-VRC-HIVMAB060-00-AB (89Zr-DFO-VRC01).
  Interventions: Drug: [89]Zr-DFO-VRC-HIVMAB060-00-AB
- Viremic HIV-infected (Experimental): Four serial PET-MR scans over 120 hours following a single, bolus injection of [89]Zr-DFO-VRC-HIVMAB060-00-AB (89Zr-DFO-VRC01).
  Interventions: Drug: [89]Zr-DFO-VRC-HIVMAB060-00-AB
- Suppressed HIV-infected (Experimental): A PET-MR scan following a single, bolus injection of [89]Zr-DFO-VRC-HIVMAB060-00-AB (89Zr-DFO-VRC01).
  Interventions: Drug: [89]Zr-DFO-VRC-HIVMAB060-00-AB

INTERVENTIONS:
Drug: [89]Zr-DFO-VRC-HIVMAB060-00-AB — Radiolabeled monoclonal antibody that targets the envelope protein of HIV-1.
  Other Names: [89]Zr-DFO-VRC01

SUMMARY:
This is a single center exploratory imaging study involving one intravenous microdose of 89Zr-DFO-VRC01 followed by whole-body PET-MR imaging in HIV infected individuals and healthy volunteers. Imaging data will be obtained from up to four static PE-MR images in order to determine dosimetry and temporal tissue uptake/tissue distribution of 89Zr-DFO-VRC01. This is not a treatment study of the biological activity of 89Zr-DFO-VRC01 to impact HIV persistence.

DETAILED DESCRIPTION:
This will be a single-center pilot study to determine dosimetry and tissue uptake/distribution and pharmacokinetics of 89Zr-VRC01. Up to 18 uninfected and HIV-infected subjects who are either taking or not taking ART will receive a small IV dose of 89Zr-VRC01. After administration of IV 89Zr-VRC01, subjects will undergo up to 4 whole body PET/MR imaging at 2, 6, 24 and 72-120h to determine the pharmacokinetics and radiation dose exposure. The study involves two phases with the second phase only to be performed only if a difference between PET activity in one or more region of interest can be determined between participant groups Phase I (HIV infected, viremic participants and healthy volunteers). Initially, up to 6 individuals with plasma HIV RNA levels >1,000 copies/ml and up to 6 HIV-uninfected individuals will be administered 89Zr radiolabeled VRC01 followed by PET-MR imaging as above (Phase 1). If differences in PET activity in one or more imaging region of interest can be identified between infected and uninfected individuals, up to 6 individuals on suppressive ART will be administered 89Zr radiolabeled VRC01 followed by PET-MRI (Phase 2). Timing of the PET-MR scans will be determined based on the data from Phase 1.

ELIGIBILITY:
Inclusion Criteria:

Study Phase 1

1. Age ≥18 years, and
2. HIV uninfected, or
3. HIV infection, and
4. has an HIV viral load measurement within 12 months of study entry of >40 copies/mL, and
5. HIV-1 envelope RNA or DNA consensus sequence from peripheral blood suggestive of VRC01 binding activity (HIV infected participants only)

Study Phase 2

1. Age ≥18 years, and
2. HIV infection, and
3. Initiated a combination ART regimen and has HIV viral load measurements below the detection limit of a clinically approved PCR-based assay (e.g. <40 HIV-1 RNA copies/mL of blood), or
4. HIV infection, and
5. has an HIV viral load measurement within 12 months of study entry of >40 copies/mL, and
6. HIV-1 envelope RNA or DNA consensus sequence from peripheral blood suggestive of VRC01 binding activity, or
7. HIV uninfected

Exclusion Criteria:

Study Phase 1

1. For patients planning to be imaged on PET-MR scanner, exclusion criteria will include any contra-indication to MRI, including permanent pacemaker, implantable metallic device/ prosthetic, aneurysm clip, non-removable piercing, or severe claustrophobia
2. Any medical condition that would compromise the imaging acquisition, in the opinion of the investigator
3. Patients who have had a study involving radiation within six months of enrolling in this study
4. Patients who are pregnant (female patients of childbearing age will be tested prior to injection of imaging agent - positive test will exclude from participating in the study)
5. Screening absolute neutrophil count <1,000 cells/mm3, platelet count <70,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <40 mL/minute, aspartate aminotransferase >100 units/L, alanine aminotransferase >100 units/L.
6. Absolute CD4+ T cell count <100 cells/μL (HIV infected individuals only)
7. Serious illness requiring hospitalization or parental antibiotics within the preceding 3 months.
8. Current HIV-related opportunistic infection such as pneumocystis pneumonia, disseminated microbacterial infection, invasive cryptococcal disease, candidal esophagitis (limited oral thrush acceptable) and cerebral toxoplasmosis

Study Phase 2

1. For patients planning to be imaged on PET-MR scanner, exclusion criteria will include any contra-indication to MRI, including permanent pacemaker, implantable metallic device/ prosthetic, aneurysm clip, non-removable piercing, or severe claustrophobia
2. Any medical condition that would compromise the imaging acquisition, in the opinion of the investigator
3. Patients who have had a study involving radiation within 12 months of enrolling in this study
4. Patients who are pregnant (female patients of childbearing age will be tested prior to injection of imaging agent - positive test will exclude from participating in the study)
5. Screening absolute neutrophil count <1,000 cells/mm3, platelet count <70,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <40 mL/minute, aspartate aminotransferase >100 units/L, alanine aminotransferase >100 units/L.
6. Absolute CD4+ T cell count <100 cells/μL (HIV infected individuals only)
7. Serious illness requiring hospitalization or parental antibiotics within the preceding 3 months.
8. Current HIV-related opportunistic infection such as pneumocystis pneumonia, disseminated microbacterial infection, invasive cryptococcal disease, candidal esophagitis (limited oral thrush acceptable) and cerebral toxoplasmosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dosimetry of 89Zr-DFO-VRC01 in healthy volunteers and HIV-infected participants. | 120 hours
  To determine the dosimetry and whole body distribution of 89Zr-DFO-VRC01 in healthy volunteers and HIV-infected participants. Study Phase 1.
89Zr-DFO-VRC01 temporal uptake in healthy controls and HIV-infected participants with viral load >1000 c/mL. | 120 hours
  To determine the differences in 89Zr-DFO-VRC01 temporal uptake in tissues in healthy volunteers versus HIV-infected, viremic participants. Study Phase 1.

SECONDARY OUTCOMES:
89Zr-DFO-VRC01 uptake in aviremic HIV-infected individuals. | 72 hours
  To evaluate the uptake and tissue distribution of 89Zr-DFO-VRC01 in HIV-infected participants on suppressive antiretroviral therapy (ART) compared with HIV-infected, viremic individuals and healthy volunteers. Study Phase 2.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henrich, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing IPD with other researchers.

REFERENCES:
- [Derived] Beckford-Vera DR, Flavell RR, Seo Y, Martinez-Ortiz E, Aslam M, Thanh C, Fehrman E, Pardons M, Kumar S, Deitchman AN, Ravanfar V, Schulte B, Wu IK, Pan T, Reeves JD, Nixon CC, Iyer NS, Torres L, Munter SE, Hyunh T, Petropoulos CJ, Hoh R, Franc BL, Gama L, Koup RA, Mascola JR, Chomont N, Deeks SG, VanBrocklin HF, Henrich TJ. First-in-human immunoPET imaging of HIV-1 infection using 89Zr-labeled VRC01 broadly neutralizing antibody. Nat Commun. 2022 Mar 9;13(1):1219. doi: 10.1038/s41467-022-28727-5. PMID 35264559